CLINICAL TRIAL: NCT01057797
Title: Nurse Managed Upper Body Strength Training in COPD
Brief Title: Nurse Managed Upper Body Strength Training in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Janet L. Larson, PhD, RN, University of Illinois at Chicago and University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NR08037
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Pulmonary rehabilitation; Self-efficacy; Muscle strength; Dyspnea; Exercise adherence
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Upper Body Strength Training with Self-Efficacy (Experimental): 16 weeks of upper body strength training combined with an exercise-specific self-efficacy enhancing intervention
  Interventions: Behavioral: Exercise-specific self-efficacy; Behavioral: upper body strength training
- Upper body strength training (Active Comparator): 16 weeks of upper body strength training with weekly health education sessions
  Interventions: Behavioral: upper body strength training
- Chair exercise (Sham Comparator): 16 wks of gentle chair exercise with weekly health education
  Interventions: Behavioral: Gentle chair exercise

INTERVENTIONS:
Behavioral: Exercise-specific self-efficacy — Subjects in the experimental group will participate in a self-efficacy enhancing intervention designed to maximize (a) exercise-specific SE-UB strength training (b) self-efficacy for overcoming barriers to exercise and (c) SE-UB physical activities. The intervention incorporates strategies to maximize the primary sources of efficacy information: (a) mastery accomplishments, (b) social modeling, (c) social persuasion, (d) interpretation of physiological and affective symptoms.
  Arms: Upper Body Strength Training with Self-Efficacy
Behavioral: Gentle chair exercise — Gentle armchair fitness exercises will be used as a sham treatment to control for the attention that subjects receive in the two strength training groups. The armchair fitness exercises will be conducted in small groups (n=8-10 per group). Armchair exercises will include stretching of all major joints with an emphasis on the arms and shoulders, massage of muscles that can be reached from the armchair (scalp, neck, shoulders, lower back, abdomen and thighs) and imagery to promote relaxation. Each session will include: 5 minutes of slow stretching, 20 minutes of faster paced exercises, 5 minutes of slower paced stretches, followed by 5-10 minutes of massage and imagery for relaxation.
  Arms: Chair exercise
Behavioral: upper body strength training — 16 weeks of lab-based upper body strength training using 8: modified lateral pull down, shoulder shrug, upright row, overhead pull down, front raise, front pull down, triceps extension, biceps curl. Training load and volume will be increased progressing from 70% to 80% of the maximum strength training and from 2 sets of 8-10 repetitions progressing to 3 sets. Each week subjects will train twice in the lab and once at home. Home exercises will include 1 set of 15-20 repetitions: biceps curl, triceps extension, front raises, lateral raises, overhead press, chest press and one-arm dumbbell row.
  Arms: Upper Body Strength Training with Self-Efficacy; Upper body strength training

SUMMARY:
This is a four month exercise training program for people with chronic obstructive pulmonary disease (COPD)with a 12 month follow-up.

DETAILED DESCRIPTION:
People with moderate to severe chronic obstructive pulmonary disease (COPD) experience intense symptoms of dyspnea when they use their arms and shoulders. To control dyspnea they avoid using their arms and ultimately experience a significant loss of upper body (UB) strength and a decrease in the level of physical activity. Some pulmonary rehabilitation programs include strength training, but the training intensity is typically very low. The purpose of this research is to examine the effects of UB strength training (designed to maximize strength gains) with a self-confidence intervention to enhance adherence to exercise. This is an experimental study with random assignment of subjects to one experimental and two control groups: (a) UB strength training and self-efficacy intervention for adherence (experimental), (b) UB strength training with health education (control 1) and (c) gentle armchair fitness exercises with health education (control 2). Each subject will be studied for a total of 16 months.The intervention period is four months in duration with a 12-month follow-up period. The sample will be people with moderate to severe COPD who experience dyspnea with UB activities. This research is innovative in that it examines the effects of upper body strength training designed to maximize strength gains and combines it with a theory-based self-efficacy (confidence-building) intervention to promote adherence to training in people with COPD.

ELIGIBILITY:
Inclusion Criteria:

* FEV1/FVC < 70 and FEV1 < 80%
* > or = 45 years of age
* Currently in stable clinical condition [free of respiratory tract infections for at least two months prior to enrollment, no recent change in the color, consistency, or quantity of sputum, afebrile and no recent change in medical therapy]
* Taking appropriate medications according to the GOLD standards
* Experience dyspnea with the use of their arms.

Exclusion Criteria:

* Evidence of restrictive lung disease or asthma
* Acute respiratory infection
* Taking oral corticosteroids on a regular basis
* >3 exacerbations in the previous year
* Evidence of significant depression (Hospital Anxiety Depression Scale >10)
* Presence of a potentially debilitating disease such as cancer, congestive heart failure, kidney disease, liver failure or cirrhosis, evidence of alcohol or drug abuse, diabetes requiring insulin therapy, musculoskeletal or degenerative nerve disease, etc.
* Presence of a condition that would make it potentially unsafe to exercise, including a history of a recent myocardial infarction, unstable angina pectoris, uncontrolled cardiac arrhythmias causing symptoms or hemodynamic compromise, severe symptomatic aortic stenosis, uncontrolled symptomatic heart failure, uncontrolled metabolic disease, abnormal response to exercise test
* Currently participating in pulmonary rehabilitation.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2003-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Upper body strength | before training, after training, 6 months post training, 12 months post training
Dyspnea | before training, after training, 6 months post training, 12 months post training
Functional performance | before training, after training, 6 months post training, 12 months post training

SECONDARY OUTCOMES:
Exercise adherence | before training, after training

CONTACTS AND LOCATIONS:
Overall Officials: Janet L Larson, PhD, RN, Principal Investigator — University of Illinois at Chicago and University of Michigan; Margaret K Covey, PhD, RN, Study Director — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Larson JL, Covey MK, Kapella MC, Alex CG, McAuley E. Self-efficacy enhancing intervention increases light physical activity in people with chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2014 Oct 3;9:1081-90. doi: 10.2147/COPD.S66846. eCollection 2014. PMID 25336939